CLINICAL TRIAL: NCT04498533
Title: Bracing or Kinesio Taping in The Management of Lateral Epicondylitis: a Randomized Single-blinded Trial
Brief Title: Bracing or Kinesio Taping in The Management of Lateral Epicondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Öznur Çelik, Principal Investigator, Haseki Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 127/29.05.2014
Record Dates: First submitted 2020-07-15; First posted 2020-08-04 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-08

CONDITIONS: Lateral Epicondylitis (Tennis Elbow)
Keywords: Lateral epicondylitis; forearm counterforce brace; kinesio taping
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Intervention Model Description: A prospective, randomized and assessor-blinded study
Who Masked: Outcomes Assessor
Masking Description: The outcome-assessing investigator (O. Celik) was blinded to the randomization. All study participants were assessed by the blinded investigator (O.Celik). Follow-up measurements were performed immediately after and one month later after treatment. All treatment sessions were applied by the same investigator (S. Sencan), who was not blinded to the study groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- B (brace) group (Active Comparator): The patients in the B group were informed about the application of the forearm strap (counterforce brace). Patients were advised to wear the counterforce brace for three weeks continuously.
  Interventions: Other: forearm strap (counterforce brace)
- KT (kinesio tape) group (Active Comparator): In the KT group, a standard 2-inch (5 cm) Kinesio®Tex tape (Kinesio Holding Corporation, Albuquerque, New Mexico, USA) was used with techniques of muscle inhibition and fascia correction. Kinesio tape was applied once a week for four weeks.
  Interventions: Other: Kinesio tape application

INTERVENTIONS:
Other: forearm strap (counterforce brace)
  Arms: B (brace) group
Other: Kinesio tape application
  Arms: KT (kinesio tape) group

SUMMARY:
Lateral epicondylitis is an overuse syndrome of the forearm, which is associated with pain and sensitivity in the lateral elbow region.

The aim of the study was to find out about is there any difference between the effects of traditional orthotic devices and adhesive taping, in the management of lateral epicondylitis. Therefore, the forearm counterforce brace, which was widely used in daily clinical practice for lateral epicondylitis, was compared with kinesio tape, a new technique of adhesive taping which has become increasingly popular. The study investigated and compared the effects of the two interventions (the forearm counterforce brace and kinesio tape) on pain severity, functional status and disability of patients with lateral epicondylitis.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 65 years
* presence of elbow pain lasting for less than three months

Exclusion Criteria:

* history of acute trauma or fracture on forearm
* congenital or acquired elbow deformities
* demyelinating diseases
* patients who had diagnosed as fibromyalgia
* presence of skin lesion on lateral aspect of the elbow
* presence of rheumatic disease
* presence of systemic infection
* presence of pregnancy
* presence of malignancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Pain Pressure Threshold | Baseline to 3 week (İmmediately after treatment)
  The tenderness on the lateral aspect of elbow was evaluated with pain pressure threshold measurements. An algometer device was used to measure pain pressure threshold. Pain pressure threshold measurements were performed at the baseline of the study, immediately after and one month later after treatment.
Grip Strength | Baseline to 3 week (İmmediately after treatment)
  Affected upper limb function was evaluated with maximal hand grip strength. Grip strength was measured with a hydraulic hand dynamometer. Grip strength was evaluated at the baseline of the study, immediately after and one month later after treatment.

SECONDARY OUTCOMES:
Patient-Rated Tennis Elbow Evaluation Questionnaire | 0 week (Baseline), 3 week (After treatment), 7 week (One month later after treatment)
  The Turkish version of Patient-Rated Tennis Elbow Evaluation Questionnaire was used in the study. Patient-Rated Tennis Elbow Evaluation Questionnaire is a 15-item self-reported questionnaire to measure perceived pain and disability in people with tennis elbow.
  The questionnaire is composed of three subscales: pain, usual activities and specific activities. Each of the items of the Patient-Rated Tennis Elbow Evaluation Questionnaire is scored on a 0-10 scale, where 0 is 'no pain' or 'no difficulty' and 10 is 'worst ever' or 'unable to do'. The total score ranges from 0 to 100, where high scores indicate greater pain and disability.
  Patient-Rated Tennis Elbow Evaluation Questionnaire was evaluated at the baseline of the study, immediately after and one month later after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Öznur Çelik, MD, Principal Investigator — University of Health Sciences, Istanbul Haseki Training and Research Hospital
Locations (1):
- University of Health Sciences, Istanbul Haseki Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Struijs PA, Smidt N, Arola H, Dijk vC, Buchbinder R, Assendelft WJ. Orthotic devices for the treatment of tennis elbow. Cochrane Database Syst Rev. 2002;(1):CD001821. doi: 10.1002/14651858.CD001821. PMID 11869609